CLINICAL TRIAL: NCT03396926
Title: Phase II Study of Pembrolizumab Plus Capecitabine and Bevacizumab in Microsatellite Stable Metastatic Colorectal Cancer
Brief Title: Pembrolizumab, Capecitabine, and Bevacizumab for Treating Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 174517; NCI-2017-02324 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Microsatellite Stable; Mismatch Repair Protein Proficient; Stage III Colorectal Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Capecitabine; Specimen Handling; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safety Lead in Cohort: Treatment (pembrolizumab, bevacizumab, capecitabine) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine PO BID on days 1-14. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Procedure: Specimen collection; Biological: Pembrolizumab
- Expansion Cohort: Treatment (pembrolizumab, bevacizumab, capecitabine) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine PO BID on days 1-14. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Procedure: Specimen collection; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Bevacizumab — Given intravenously (IV)
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Capecitabine — Given orally (PO)
  Other Names: Ro 09-1978/000; Xeloda
Procedure: Specimen collection — For use in correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the side effects and best dose of capecitabine when given together with pembrolizumab and bevacizumab, and investigates how well they work in treating patients with microsatellite stable colorectal cancer that has spread to nearby tissues or lymph nodes, has spread to other places in the body, or that cannot be removed by surgery. Monoclonal antibodies, such as pembrolizumab and bevacizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving capecitabine together with pembrolizumab and bevacizumab may work better in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D)/maximum tolerated dose (MTD) of capecitabine when administered with pembrolizumab and bevacizumab. (Safety Lead-In Cohort) II. To evaluate the overall response rate (ORR) to pembrolizumab plus capecitabine and bevacizumab (complete or partial response rate per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) in subjects with metastatic or locally advanced unresectable microsatellite stable (MSS)/mismatch repair proficient (pMMR) colorectal carcinoma (CRC) that is stable or progressing on fluorouracil (5FU)-based therapy. (Phase II Expansion Cohort)

SECONDARY OBJECTIVES (Phase II Expansion Cohort):

I. To determine the safety and tolerability of pembrolizumab in combination with capecitabine and bevacizumab.

II. To evaluate ORR per immune-related RECIST (irRECIST). III. To evaluate duration of response (DOR), disease control rate (DCR) and progression-free survival (PFS) per RECIST 1.1 and irRECIST and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Correlation of outcomes to line of therapy; stable disease or progression on a prior regimen containing infusional 5-FU or capecitabine; prior exposure to bevacizumab; and primary tumor location.

II. To explore baseline immune profiles via PD-L1, and multiplex Immunohistochemistry (IHC) for identification of potentially predictive biomarkers in patients with metastatic or locally advanced, unresectable CRC treated with pembrolizumab-based combination therapy.

III. To characterize the change in the populations of tumor-infiltrating immune cells (TIICs) by IHC induced by pembrolizumab-based combination therapy in paired pre- and on-treatment tumor biopsies from patients with metastatic or locally advanced, unresectable MSS / pMMR CRC.

IV. To determine the change in T cell repertoire via next generation sequencing (NGS) within blood and tumor biopsy samples induced by pembrolizumab-based combination therapy in patients with metastatic or locally advanced, unresectable MSS/pMMR CRC.

V. To establish human immune system (HIS) patient-derived xenograft (PDX) models from pre-treatment biopsies to a) analyze change in immune cell profiles HIS PDX models using the same techniques as described for corresponding patients, above and b) correlate response to pembrolizumab-containing therapy in patients and HIS PDX.

OUTLINE:

An initial safety lead-in will be performed to define the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D). Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine orally (PO) twice daily (BID) on days 1-14. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 9 weeks until disease progression, start of new anti-cancer therapy, death, or end of the study whichever comes first

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed, locally advanced unresectable or metastatic (stage IV) colorectal adenocarcinoma
2. Have locally confirmed MSS or pMMR CRC; MSS is defined as 0-1 allelic shifts among 3-5 tumor microsatellite loci using a PCR-based assay; pMMR is defined as presence of protein expression of 4 MMR enzymes (DNA mismatch repair protein Mlh1 (MLH1), DNA mismatch repair protein Msh2 (MSH2), mutS homolog 6 (MSH6) and Mismatch repair endonuclease postmeiotic segregation increased 2 (PMS2) by immunohistochemistry.
3. Have stable disease or progression on a prior regimen containing infusional 5-FU or capecitabine according to the interpretation of the treating provider
4. Be willing and able to provide written informed consent/assent for the trial
5. Be 18 years of age on day of signing informed consent
6. Have measurable disease based on RECIST 1.1
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion (phase II dose expansion cohort only); newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1; subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor
8. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
9. Demonstrate adequate organ function performed within 10 days of treatment initiation as defined below:

   1. Absolute neutrophil count (ANC) >= 1,500 /mcL
   2. Platelets >= 100,000 / microliter (mcL)
   3. Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
   4. Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN. Glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)). Creatinine clearance should be calculated per institutional standard
   5. Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN. Patients with Gilbert's disease may be included if their direct bilirubin is ≤ 1.5 X ULN.
   6. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT)) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
   7. Albumin >= 2.5 mg/dL
   8. International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   9. Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy; as long as PT or PTT is within therapeutic range of intended use of anticoagulants
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
11. Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication
12. Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy

    * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
3. Has a known history of active tuberculosis (TB) (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients
5. Hypersensitivity/intolerance to capecitabine, Infusional 5-Fluorouracil (5-FU), or bevacizumab
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

   * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
8. Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
11. Has known history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
12. Has an active infection at the time of cycle 1 day 1 requiring systemic therapy
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
17. Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
18. Has known active hepatitis B (e.g., hepatitis B surface antigen (HBsAg) reactive) or hepatitis C (e.g., hepatitis C virus (HCV) ribonucleic acid [RNA] [qualitative] is detected)
19. Requires therapeutic anticoagulation with warfarin at baseline. Patients must be off warfarin or warfarin-derivative anti-coagulants for at least 7 days prior to starting study drug, however, therapeutic or prophylactic therapy with low-molecular weight heparin is allowed
20. Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug
21. Known bleeding risk including serious hemorrhage or hemoptysis within the last 3 months; major surgery within the past 8 weeks or minor surgery within the past 4 weeks
22. Has known gastrointestinal bleeding or any other hemorrhage/bleeding event Common Terminology Criteria for Adverse Events (CTCAE) grade > 3 within 6 months of start of study drug
23. Has greater than 1+ proteinuria on a urine dipstick or equivalent routine laboratory analysis will require further testing with a urine protein to creatinine ratio (UPCR); UPCR must be calculated as follows: UPCR = protein concentration (mg/dL)/creatinine (mg/dL); if the UPCR >= 1, then the patient will not be eligible for study entry; however, if urinalysis or equivalent routine laboratory analysis shows no protein, then UPCR testing is not required
24. Has a history of non-healing wounds or ulcers, or bone re-fractures within 3 months of fracture
25. Has a history of arterial thromboembolism within 12 months of start of study drug
26. Has inadequately controlled hypertension (defined as systolic blood pressure greater than 150 mm Hg or diastolic blood pressure greater than 95 mm Hg). The use of anti-hypertensive medications to control blood pressure is permitted. Retesting is permitted.
27. Has a history of hypertensive crisis or hypertensive encephalopathy within 6 months prior to planned start of study drug
28. Has had clinically significant cardiovascular disease within 12 months of planned start of study drug, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication, percutaneous transluminal coronary angioplasty/stent
29. Has a known history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to planned start of study drug
30. Known reversible posterior leukoencephalopathy syndrome (RPLS)
31. Difficulty swallowing, malabsorption, active partial or complete bowel obstruction, or other chronic gastrointestinal disease or conditions that may hamper compliance and/or absorption of capecitabine
32. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chloe Atreya, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in safety lead in cohort will be included in expansion cohort as All Subjects as Treated (ASaT) population. ASaT population will be used for analysis of objective response (ORR), disease control (DCR), progression-free survival (PFS) and overall survival (OS) and consist of participants who received at least one dose of study treatment (200mg pembrolizumab, 7.5mg/kg bevacizumab and 1000mg/m2 capecitabine). Participants ineligible for safety analysis will be replaced.
Groups:
- Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine); Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine): Participants received 200 mg pembrolizumab IV over 30 minutes on day 1, 7.5 mg/kg bevacizumab IV over 30-90 minutes on day 1, and 1000 mg/m2 capecitabine orally (PO) twice a day (BID) on days 1-14. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.
Period: Safety Lead In Cohort
Arm/Group | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) | Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine)
Started | 7 | 0
Completed | 6 (One participant was deemed ineligible for safety analysis but was included in the ASaT analyses.) | 0
Not Completed | 1 | 0
Period: Expansion Cohort
Arm/Group | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) | Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine)
Started | 7 | 37
Completed | 7 | 33
Not Completed | 0 | 4
Not completed — Participants did not complete follow-up scan required for disease response outcomes | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine): Participants receive pembrolizumab IV over 30 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine orally (PO) twice a day (BID) on days 1-14. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) | Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) | Total
Number analyzed (Participants) | 7 | 37 | 44
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 0 | 1 | 1
  30-39 years old | 2 | 7 | 9
  40-49 years old | 0 | 7 | 7
  50-59 years old | 4 | 11 | 15
  60-69 years old | 1 | 7 | 8
  70-79 years old | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 19 | 22
  Male | 4 | 18 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 6 | 27 | 33
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 5 | 25 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 37 | 44

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment-related, Dose-limiting Toxicities (DLT) (Safety Lead-In Cohort)
Description: A DLT evaluation of the first 6 participants will be conducted to confirm the safety of administering pembrolizumab at 200 mg (flat dosing) every three weeks with capecitabine and bevacizumab and include all participants in the safety lead in cohort who received at least 1 dose of study treatment. At least one laboratory or vital sign measurement obtained subsequent to at least one dose of study treatment is required for inclusion in the analysis including a baseline measure. Dose-limiting toxicity (DLT) must be clinically-significant toxicities which are at least possibly treatment-related per the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4
Time Frame: Up to 1 cycle (each cycle is 21 days)
Measure: Number; unit: proportion of participants
Arm/Group | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine)
Number analyzed (Participants) | 6
proportion of participants | 0.33

2. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of the participants in the ASaT population who have a confirmed complete response (CR) or a partial response (PR) (Overall Response (OR) = CR + PR) assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 on Computerized Tomography (CT) or magnetic resonance imaging or (MRI) imaging if a CT cannot be obtained. The ORR and 95% confidence interval will be provided using exact binomial method proposed by Clopper and Pearson (1934).
Time Frame: Up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ASaT Population (Pembrolizumab, Bevacizumab, Capecitabine): All participants who received pembrolizumab IV over 30 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, and capecitabine PO BID on days 1-14. Treatment repeats every 3 weeks for up to 35 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | ASaT Population (Pembrolizumab, Bevacizumab, Capecitabine)
Number analyzed (Participants) | 40
percentage of participants | 5 [0.6 to 16.9]

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who have achieved confirmed CR or PR or have demonstrated stable disease (SD) for at least 24 weeks prior to any evidence of progression assessed by RECIST and immune-related RECIST (irRECIST). The percentage of participants and 95% confidence interval, will be provided using exact binomial method proposed by Clopper and Pearson (1934).
Time Frame: Up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ASaT Population (Pembrolizumab, Bevacizumab, Capecitabine)
Number analyzed (Participants) | 40
percentage of participants | 25 [16.7 to 41.2]

4. Secondary Outcome: Median Duration of Response (DOR)
Description: Duration of response is defined as the time from first documented evidence of CR or PR assessed by RECIST and irRECIST until disease progression or death due to any cause, whichever occurs first. Kaplan-Meier (KM) curves and median estimates from will be reported
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASaT Population (Pembrolizumab, Bevacizumab, Capecitabine)
Number analyzed (Participants) | 40
months | 13.5 [12.3 to NA] — The upper range of the confidence interval was calculated to be infinity

5. Secondary Outcome: Median Overall Survival (OS)
Description: OS is defined as the time from first day of study treatment to death due to any cause. Subjects without documented death at the time of the final analysis will be censored at the date of the last follow-up. KM curves and median estimates from the KM curves will be provided as appropriate.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASaT Population (Pembrolizumab, Bevacizumab, Capecitabine)
Number analyzed (Participants) | 40
months | 10.1 [8.52 to 15.2]

6. Secondary Outcome: Median Progression-Free Survival (PFS)
Description: PFS is defined as the time from first day of study treatment to the first documented disease progression or death due to any cause, whichever occurs first. Median estimates in months and the 95% confidence interval will be reported.
Time Frame: Up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ASaT Population (Pembrolizumab, Bevacizumab, Capecitabine)
Number analyzed (Participants) | 40
months | 4.29 [3.68 to 6.05]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) | Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine)
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/37
Serious Adverse Events (participants affected / at risk) | 4/7 | 11/37
Other Adverse Events (participants affected / at risk) | 7/7 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) (N=7) | Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) (N=37)
Abdominal pain (Gastrointestinal disorders) | 2 (7) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) — Pneumoperitoneum
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) — Failure to thrive
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0) — Systemic Inflammatory Response Syndrome
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) — Pulmonary embolism
Urinary tract pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead in Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) (N=7) | Expansion Cohort: Treatment (Pembrolizumab, Bevacizumab, Capecitabine) (N=37)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 18 (26)
Nausea (Gastrointestinal disorders) | 4 (13) | 13 (17)
Constipation (Gastrointestinal disorders) | 1 (2) | 15 (17)
Diarrhea (Gastrointestinal disorders) | 4 (7) | 10 (13)
Mucositis oral (Gastrointestinal disorders) | 4 (12) | 10 (17)
Vomiting (Gastrointestinal disorders) | 3 (8) | 10 (16)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (5)
Oral pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 5 (11) | 24 (29)
Non-cardiac chest pain (General disorders) | 2 (2) | 8 (10)
Fever (General disorders) | 3 (5) | 5 (9)
Edema limbs (General disorders) | 1 (3) | 5 (6)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 4 (4)
Chills (General disorders) | 1 (2) | 4 (5)
Flu like symptoms (General disorders) | 1 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (20) | 20 (61)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (9) | 10 (11)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3) | 10 (12)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (12) | 6 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 8 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (8) | 14 (30)
Weight loss (Investigations) | 4 (12) | 9 (16)
Aspartate aminotransferase increased (Investigations) | 1 (3) | 7 (8)
Platelet count decreased (Investigations) | 1 (1) | 7 (18)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5)
Weight gain (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (3)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 9 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 6 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (10) | 13 (15)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (8) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (9)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 8 (14)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 3 (4)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (2)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (7) | 7 (8)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (8) | 5 (6)
Dizziness (Nervous system disorders) | 1 (2) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (4) | 1 (2)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 5 (11)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (4) | 3 (3)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (6) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03396926/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT03396926/ICF_001.pdf